CLINICAL TRIAL: NCT06396572
Title: Enhancing Clinical Procedures Through Deliberate Practice Using Immersive Virtual Reality
Brief Title: Immersive Virtual Reality (IVR) Procedure
Acronym: IVR-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Lau Siew Tiang, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IVR-Procedure
Record Dates: First submitted 2024-04-15; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Procedure
Keywords: urinary catheterisation; Immersive Virtual Reality; Clinical competency; Clinical procedures; Nursing

STUDY DESIGN:
Intervention Model Description: Cluster randomization trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality (Experimental): The Participants used Immersive Virtual Reality for learning and practice urinary catheterisation procedure
  Interventions: Procedure: IVR-Procedure
- Nursing clinical laboratory (Active Comparator): The Participants used a traditional nursing clinical laboratory for face to face learning and practice urinary catheterisation procedure
  Interventions: Procedure: Nursing Clinical Laboratory practice

INTERVENTIONS:
Procedure: IVR-Procedure — Using immersive virtual reality to learn urinary catheterisation procedure
  Arms: Immersive Virtual Reality
Procedure: Nursing Clinical Laboratory practice — Using nursing clinical laboratory sessions to learn urinary catheterisation procedure
  Other Names: Active Comparator
  Arms: Nursing clinical laboratory

SUMMARY:
A pilot randomised controlled trial to assess the nursing students' learning outcomes of the urinary catheterisation procedure by comparing the immersive virtual reality (IVR) to traditional lab sessions.

DETAILED DESCRIPTION:
Design: A pilot randomised controlled trial was employed to assess the learning outcomes of the urinary catheterisation procedure by comparing the immersive virtual reality (IVR) intervention to traditional lab sessions.

Eligibility: Second-year undergraduate nursing students (n = 200) enrolled into the module NUR2125 (Pathophysiology, Pharmacology and Nursing Practice II) were invited to participate in the study.

Setting: The study was conducted at a university in Singapore from January to April 2023.

Procedure: Ten lab groups of second-year undergraduate nursing students were invited to participate in the study. They received the standard blended learning activities, which included clinical lab sessions and videos on the urinary catheterisation procedure. Out of the ten groups, four groups were randomly allocated to the IVR intervention group, and another four groups were randomly assigned to the waitlist control group (traditional lab sessions).

1. For the intervention group (IVR), the students used the IVR device for practice in class under the supervision of their tutor. They then loaned the IVR device for two weeks for home practice.
2. For the waitlist control group (traditional lab sessions), they learned and practiced the urinary catheterisation procedure in class. Students received the additional intervention (using the IVR device for home practice) after the collection of post-test data.

Data collection: Prior to lab practice, each participant completed a demographic survey and a set of pre-test questionnaires on personality inventory, cognitive load, and representation of VR in education. Only students who voluntarily joined the programme were recruited into the study.

The participants completed the post-test questionnaires in March 2023 prior to their formative clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Year 2 Nursing students enrolled in the PPNP2 module

Exclusion Criteria:

* Students who declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Cognitive Load | 3 months
  The Cognitive Load Scale (CLS) was adapted from Leppink et al. (2013) and analyses the level of working memory resources needed to process information. It consists of 10 items that are rated on an 11-point scale (0 = Not at all the case to 10 = Completely the case). Items 1 to 3 relate to intrinsic load, items 4 to 6 fall under extraneous load, and items 7 to 10 are associated with germane load. Responses are added to give a total score for each subscale, which ranges from 0 (lowest) to 30 or 40 (highest) in the case of the germane load subscale. Higher total scores indicate more working memory resources required to process the information load under different conditions.

SECONDARY OUTCOMES:
Clinical skill competency | 3 months
  To evaluate the skills competency, the nursing students were assessed by their tutors using a competency assessment tool based on the skills checklist. Within the checklist, it determined the performance of the participants on completing the procedural steps on a 10-point scale (0-3 = Need improvement, 4-6 = Meet expectation, 7-9 = Exceed expectation), which was computed into a percentage score. Higher scores indicate a higher competency level in conducting the urinary catheterization procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Tiang LAU, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Alice Lee Centre for Nursing Studies, Singapore, Singapore